CLINICAL TRIAL: NCT03232515
Title: The Use of Electrical Bioimpedance to Evaluate Dry Weight in Patients With Chronic Renal Failure in Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Sonora (Other)
Responsible Party: Principal Investigator, Mauro Eduardo Valencia Juillerat, P.H.D. Principal researcher, Universidad de Sonora
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DMCS/CBIDMCS/D-87bis
Record Dates: First submitted 2017-07-14; First posted 2017-07-28 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Chronic Renal Failure; Dialysis; Dry Weight; Blood Pressure
Keywords: Bioimpedance Vector Analysis (BIVA); Chronic Renal Failure; Dialysis; Dry weight; Blood Pressure
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Non-randomized pre-test / post-test clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Evaluation,estimation and modification of the dry weight by BIVA.
  Interventions: Combination Product: To estimate the dry weight of patients with chronic renal failure under hemodialysis treatment using BIVA

INTERVENTIONS:
Combination Product: To estimate the dry weight of patients with chronic renal failure under hemodialysis treatment using BIVA — Using the BIVA method, excess fluid will be estimated in patients with chronic renal failure undergoing hemodialysis in order to obtain a better estimate of dry weight and thus improve the quality of life of patients.

SUMMARY:
INTRODUCTION: Accurate estimation of dry weight (DW) is an important and difficult problem in clinical practice. DW is defined as the lowest weight after hemodialysis (HD) where the patient will not develop symptoms of hypotension and edema, in addition to not using antihypertensives. Achieving a fluid balance benefits the control of blood pressure and reduces cardiovascular risk. In most HD centers, the DW is estimated using a subjective method dependent on the signs and symptoms that the patient presents. Recently, several approaches have been studied to develop a standardized DW evaluation technique. Among these, the analysis of electric bioimpedance vectors (BIVA) has been recognized as a simple and promising method with high reproducibility.

OBJECTIVE: To use BIVA to improve dry weight estimation in patients with chronic renal failure undergoing hemodialysis.

Methods: This is a non-randomized pre-test / post-test clinical trial, where the universe of patients comes from the hemodialysis unit of the General State Hospital of Sonora.

Patients who have limb amputations, pacemakers, metal implants, who are under renal transplant protocol or who have a renal transplant, and presence of infectious foci will be restricted from participating.

The diagnosis of DW in the patients will be performed for modification and follow-up. Fluid status will be evaluated using BIVA. Measurements will be made before and after HD in three consecutive weekly periods and one one final assessment at three months.

At the beginning of each period, weight, electrolytes, creatinine, total proteins, albumin, pre-albumin, urea and blood pressure will be measured to calculate the Malnutrition Inflammation Score and Bilbrey Index. At the end of the HD protocol of each period, body composition and muscle strength will be evaluated through triceps skinfold, mid-upper arm circumference and dynamometry. The dialysis dose received will be modified according to BIVA.

The main variables to be considered will be DW, extracellular water and blood pressure.

The duration of the study will be approximately 6 months. In addition, at the end of each measurement, each participant will be given a nutritional recommendation (feeding guide) specific to their energy requirements.

DETAILED DESCRIPTION:
* Place of study: General Hospital of the State of Sonora "Dr. Ernesto Ramos Bours" in the city of Hermosillo, Sonora.
* Sociodemographic and symptomatological information questionnaire: Questionnaires will be applied to each participant, which will allow to obtain information of their occupation, residence, date of birth, their own medical and family history, as well as typical symptoms of the diseases.
* Weight: The weight will be measured with a SECA Model 813 Portable Floor Scale. The person should wear light clothing, empty pockets, without shoes, accessories (belts, necklaces, watches, etc.); In a firm position, facing forward, without movement at the time of taking the measurement. Weight measurement should be the simplest and most accurate of anthropometric measurements, the balance should be calibrated periodically.
* Height: The height will be measured with a portable stadiometer Model 217 SECA. The participant is presented for the measurement of the height dressed with the minimum of clothes, at least, without shoes and socks. The participant is instructed to stand on the stadiometer so that his heels, gluteus, and shoulder blades are in contact with the back plate, and the heels together. The head should be placed on the "Frankfurt Plane", the head of the instrument will move down to make contact with the apex of the skull. With the subject in the correct position, he is instructed: "take a deep breath and stand tall". The height is measured at the point of inspiration without pressure being applied.
* Single-frequency bioimpedance (BIA): The BIA measurement will be performed according to the established criteria by the National Institute of Health Technology Assessment Conference Statement. The subject will be placed supine, with arms and legs separated from the body and palms down. The electrodes will be located in the right extremities, located on the back of the hand and foot near the phalangeal-metacarpal and phalangeal-metatarsal joints and in the styloid process of the wrist and between the medial and lateral malleolus of the ankle, through which an imperceptible electric current will be introduced.

The subjects should be under the following conditions so that the study can be carried out:

* Fast four hours before the measurement.
* Not having consumed alcoholic beverages during the 48 hours prior to the test.
* No strenuous exercise 24 hours prior to measurement.
* In the case of women, do not menstruate.
* Do not have any metal objects on the body.
* The approximate measurement time is five minutes.

  * Vector analysis of electric bioimpedance (BIVA): The variables of resistance (R), Reactance (Xc) and size of each of the individuals measured to be plotted in the reference ellipses of the Mexican population by sex will be used. The R and Xc standardized by size (R / size and Xc / size) will be used to plot the vector of individuals within the percentiles 50, 75 and 95% of tolerance ellipses, differentiated by sex, using the BIVA program Software 2002.
  * Clinical assessment of dry weight and hemodialysis (HD) process: Based on the traditional practices of the Hospital dialysis unit, the physician / nurse will perform physical examination and interpret the signs and symptoms associated with the renal disease, these are blood pressure , heart rate, respiratory rate, temperature, presence of infection and edema. This will include present and past health-disease aspects, medications, as well as information on the patient's daily life. Upon arrival, the patient will be weighed according to the methodology described above. According to the traditional practice of the Hospital Dialysis Unit, the patient's target weight will be based on the difference between the post-dialysis weight of the last session and the current weight, in addition to taking into account the signs and symptoms Mentioned above, In order to determine the excess water of the patient.

The amount of fluid to be withdrawn to the patient, the ultrafiltration rate and the duration time are determined by the nephrologist physician in consultation prior to the HD session. Such information may be modified in the HD session depending on the clinical evaluation of the patient on the day of treatment.

Before starting HD, the patient's vascular access is prepared with three alcohol times and three times of 10% EXSEPT, and the clot is removed from the access.

The time, ultrafiltration rate and the amount of liquid to be filtered on the HD machine (Fresenius Medical Care 4008 S - OCM Kt / V) are then programmed. Once programmed, it connects To the patient and heparin is administered at an initial bolus and at each hour of treatment. A total of 100 units per kg of body weight is given and the total is divided between the initial bolus and each hour of treatment. The mechanism by which the HD machine works is as follows: A pump directs the patient's blood to a filter of Polysulfone fibers, blood runs up-down, while a dialysing solution (its content is similar to normal blood plasma) flows in the opposite direction. By means of osmosis and the pressure exerted by the filter, excess substances are removed from the patient's blood and, if any of the plasma components are deficient, is absorbed from the dialysing solution. The blood is returned to the patient and heparin is supplied at both catheter outlets to avoid coagulation. The catheter is then sealed with a stopper and a patch is placed to prevent contact with the outside medium. Finally, the vital signs are reviewed again and the appointment is scheduled for the next treatment. In case the vital signs are altered, the patient is immediately referred to the emergency department.

* Laboratory parameters: Pre and post-dialysis patient blood samples will be taken to analyze the following parameters: serum electrolytes, blood biometrics, blood chemistry and Hepatic function. If feasible, the PCR will be analyzed.
* Blood pressure: Blood pressure will be measured with an automatic monitor included in the hemodialysis equipment (Fresenius Medical Care 4008 S - OCM Kt / V). To perform the measurement, the patient has to be relaxed and seated comfortably, at a comfortable ambient temperature. Do not bathe, drink alcohol or caffeine, smoke, exercise or eat 30 minutes before taking the measurement. The participants should sit in a chair with their feet flat on the floor, the back straight and the arm band should be at the same level as their heart with the palm up and relaxed. The nurse will start by palpating the arm for the pulse of the brachial artery, where the diaphragm of the stethoscope will be placed. This artery is located between the brachial and brachial biceps muscles; In its lower-lateral path accompanies the median nerve. The bracelet should be placed to take the measurement.Special considerations: - In patients with peripheral insertion of central catheters, the upper arm should be avoided in which there is a central peripheral insertion catheter. - In patients with a bypass Dialysis, or fistula, blood pressure should be taken in the opposite arm if the patient has an arteriovenous insertion or fistula necessary for dialysis, this is to avoid possible trauma or clot formation.
* Nutritional intervention: Patients will be made aware of the importance of adherence to nutritional treatment through individualized sessions, addressing the following topics: a) how to ensure adequate energy and protein intake, b) how to control fluid, sodium and potassium intake, identifying foods rich in them, c) Incorrect feeding, d) food preparation techniques, among others. Also, in each session, depending on the patient's nutritional status, laboratory values and comorbidities, a personalized feeding guide will be provided, which will include the foods to be consumed and in what quantities, using the Mexican equivalents system for renal patients and the current Kidney Disease Improving Global Outcomes (KDIGO) practice guidelines.
* Malnutrition Inflammation Score (MIS), Bilbrey Index and subjective global assessment: These are instruments that will be used to establish a Nutritional diagnosis of each patient. Clinical, biochemical and anthropometric parameters are evaluated. Each of the measurements will be made according to the current standardized methodology.

ELIGIBILITY:
Inclusion Criteria:

* Must be patient of the Hospital
* Diagnosed with chronic renal failure (KDOQI stage 5)
* >18 years
* Undergoing Hemodialysis treatment

Exclusion Criteria:

* Amputations
* Have metalic implants
* Have pacemaker
* Renal transplant (or in protocol to receive it)
* Infectious processes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2018-02-07 (Actual); Study Completion 2018-08-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Systolic Blood Pressure at 6 months | 6 months
  (mm Hg)
Change from Baseline Dry weight at 6 months | 6 months
  (Kg)

SECONDARY OUTCOMES:
Height | 6 months
  Meters
Change from Baseline Tricep skinfold at 6 months | 6 months
  mm
Elbow width | 6 months
  cm
Change from Baseline Arm circumference at 6 months | 6 months
  cm
Change from Baseline Dynamometry at 6 months | 6 months
  Kg
Change from Baseline Seric glucose at 6 months | 6 months
  mg/dL
Change from Baseline Seric cholesterol at 6 months | 6 months
  mg/dL
Change from Baseline Seric creatinine at 6 months | 6 months
  mg/dL
Change from Baseline Total proteins at 6 months | 6 months
  g/dL
Change from Baseline Albumin at 6 months | 6 months
  mg/dL
Change from Baseline Pre-albumin at 6 months | 6 months
  mg/dL
Change from Baseline Blood urea nitrogen at 6 months | 6 months
  mg/dL
Change from Baseline Reactive C protein at 6 months | 6 months
  mg/L
Change from Baseline Chloride at 6 months | 6 months
  meq/L
Sodium | 6 months
  meq/L
Change from Baseline Potassium at 6 months | 6 months
  meq/L
Change from Baseline Calcium at 6 months | 6 months
  mg/dL
Change from Baseline Magnesium at 6 months | 6 months
  mg/dL
Change from Baseline Phosphorus at 6 months | 6 months
  mg/dL
Change from Baseline Transferrin at 6 months | 6 months
  mg/dL
Change from Baseline Lymphocytes at 6 months | 6 months
Change from Baseline Leukocytes at 6 months | 6 months
  (10^3)/uL
Change from Baseline Single frequency bioimpedance at 6 months | 6 months
  Resistance and Reactance
Change from Baseline Nutritional Status at 6 months | 6 months
  Bilbrey Index (BI)
Change from Baseline Extracellular water at 6 months | 6 months
  (Liters)
Change from Baseline Nutritional Status at 6 months | 6 months
  Subjective Global Assessment (SGA)
Change from Baseline Nutritional Status at 6 months | 6 months
  Malnutrition-Inflammation Score (MIS)

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Eduardo Valencia Juillerat, P.H.D., Principal Investigator — Universidad de Sonora
Locations (1):
- Hospital General del Estado de Sonora "Dr. Ernesto Ramos Bours", Hermosillo, Sonora, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lavilla Royo FJ. Protocolo diagnóstico de los edemas. Medicine 10(79):5379-82, 2011.
- [Background] Bekheirnia MR, Schrier RW. Pathophysiology of water and sodium retention: edematous states with normal kidney function. Curr Opin Pharmacol. 2006 Apr;6(2):202-7. doi: 10.1016/j.coph.2005.09.008. Epub 2006 Feb 17. PMID 16483846
- [Background] Chaney E, Shaw A. Pathophysiology of fluid retention in heart failure. Contrib Nephrol. 2010;164:46-53. doi: 10.1159/000313720. Epub 2010 Apr 20. PMID 20427993
- [Background] Koomans HA. Pathophysiology of oedema in idiopathic nephrotic syndrome. Nephrol Dial Transplant. 2003 Aug;18 Suppl 6:vi30-2. doi: 10.1093/ndt/gfg1063. PMID 12953039
- [Background] Muldoon J. Assessment and monitoring of oedema. Journal of Community Nursing. November/December 2011, volume 25, issue 6.
- [Background] Trayes KP, Studdiford JS, Pickle S, Tully AS. Edema: diagnosis and management. Am Fam Physician. 2013 Jul 15;88(2):102-10. PMID 23939641
- [Background] Casey G. Oedema: causes, physiology and nursing management. Nurs Stand. 2004 Sep 1-7;18(51):45-51; quiz 52. doi: 10.7748/ns.18.51.45.s54. PMID 15487497
- [Background] Cameron N. Essential anthropometry: Baseline anthropometric methods for human biologists in laboratory and field situations. Am J Hum Biol. 2013 May-Jun;25(3):291-9. doi: 10.1002/ajhb.22388. No abstract available. PMID 23606226
- [Background] National Institute for Health and Care Excellence (NICE). The BCM - Body Composition Monitor for managing fluid in people having dialysis. Medtech innovation briefing. Published: 13 October 2015
- [Background] Frese EM, Fick A, Sadowsky HS. Blood pressure measurement guidelines for physical therapists. Cardiopulm Phys Ther J. 2011 Jun;22(2):5-12. PMID 21637392
- [Background] Perez Lizaur, Palacios González. Sistema Mexicano de Equivalentes para Paciente Renal. Fomento de Nutrición y Salud. México D.F, julio 2009
- [Background] Piccoli A, Nescolarde LD, Rosell J. [Conventional and vectorial analysis of bioimpedance in clinical practice]. Nefrologia. 2002;22(3):228-38. No abstract available. Spanish. PMID 12123122
- [Background] NIH Consensus statement. Bioelectrical impedance analysis in body composition measurement. National Institutes of Health Technology Assessment Conference Statement. December 12-14, 1994. Nutrition. 1996 Nov-Dec;12(11-12):749-62. PMID 8974099
- [Result] Jian Y, Li X, Cheng X, Chen Y, Liu L, Tao Z, Zuo L. Comparison of bioimpedance and clinical methods for dry weight prediction in maintenance hemodialysis patients. Blood Purif. 2014;37(3):214-20. doi: 10.1159/000362109. Epub 2014 Jun 5. PMID 24902760
- [Result] Hyun SH, Choi JY, Cho JH, Park SH, Kim CD, Kim YL. Assessment of fluid and nutritional status using multifrequency bioelectrical impedance analysis in peritoneal dialysis patients. Blood Purif. 2014;37(2):152-62. doi: 10.1159/000360272. Epub 2014 Apr 26. PMID 24777057
- [Result] Stevens PE, Levin A; Kidney Disease: Improving Global Outcomes Chronic Kidney Disease Guideline Development Work Group Members. Evaluation and management of chronic kidney disease: synopsis of the kidney disease: improving global outcomes 2012 clinical practice guideline. Ann Intern Med. 2013 Jun 4;158(11):825-30. doi: 10.7326/0003-4819-158-11-201306040-00007. PMID 23732715
- [Result] Atilano-Carsi X, Miguel JL, Martinez Ara J, Sanchez Villanueva R, Gonzalez Garcia E, Selgas Gutierrez R. [Bioimpedance vector analysis as a tool for the determination and adjustment of dry weight in patients undergoing hemodialysis]. Nutr Hosp. 2015 May 1;31(5):2220-9. doi: 10.3305/nh.2015.31.5.8649. Spanish. PMID 25929397
- [Result] Espinosa-Cuevas Mde L, Rivas-Rodriguez L, Gonzalez-Medina EC, Atilano-Carsi X, Miranda-Alatriste P, Correa-Rotter R. [Bioimpedance vector analysis for body composition in Mexican population]. Rev Invest Clin. 2007 Jan-Feb;59(1):15-24. Spanish. PMID 17569296
- [Result] Espinosa Cuevas MA, Navarrete Rodriguez G, Villeda Martinez ME, Atilano Carsi X, Miranda Alatriste P, Tostado Gutierrez T, Correa-Rotter R. Body fluid volume and nutritional status in hemodialysis: vector bioelectric impedance analysis. Clin Nephrol. 2010 Apr;73(4):300-8. PMID 20353738
- [Result] Gonzalez-Ortiz AJ, Arce-Santander CV, Vega-Vega O, Correa-Rotter R, Espinosa-Cuevas Mde L. Assessment of the reliability and consistency of the "malnutrition inflammation score" (MIS) in Mexican adults with chronic kidney disease for diagnosis of protein-energy wasting syndrome (PEW). Nutr Hosp. 2014 Oct 4;31(3):1352-8. doi: 10.3305/nh.2015.31.3.8173. PMID 25726233
- See also: The National Kidney Foundation produces clinical practice guidelines through the NKF Kidney Disease Outcomes Quality Initiative (NKF KDOQI)™. This program has provided evidence-based guidelines for all stages of chronic kidney disease (CKD) — https://www.kidney.org/professionals/guidelines